CLINICAL TRIAL: NCT03958786
Title: Frailty in People Living With HIV Aged 70 Years or More : Screening Feasibility, Prevalence, Risk Factors and Impact on Pejorative Events
Brief Title: Frailty in People Living With HIV Aged 70 Years or More
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ANRS EP66 SEPTAVIH
Record Dates: First submitted 2019-05-20; First posted 2019-05-22 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: Multicenter, prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): 500 HIV-1 infected patients, aged 70 years and older
  Interventions: Other: Simplified Geriatric Evaluation; Other: Sampling

INTERVENTIONS:
Other: Simplified Geriatric Evaluation — * Questionnaires
  * Self assessment questionnaires
  * Mobility and balance tests
Other: Sampling — - Blood samples : 35 ml will be collected at baseline, after signature of written informed consent, 7 ml at M12

SUMMARY:
The ANRS EP66 SEPTAVIH Study aims to screen feasibility of evaluating frailty in people living with HIV aged 70 or older, to estimate its prevalence, to analyse associated risk factors and to evaluate the impact of frailty on pejorative events.

SEPTAVIH is a French, multicentre, prospective, observational study which will include 500 HIV-infected participants

DETAILED DESCRIPTION:
The primary objective is to assess the prevalence of frailty at baseline in People living with HIV (PLWH) aged 70 years and older, using the Fried index.

The main secondary objectives of this study are :

* To assess frequency frailty according to different indexes or scores (Fried, Health deficits Index, HAS score, VACS index)
* To evaluate the association between frailty and specific HIV-related characteristics (for example known duration of HIV infection), or non-specific factors (such as non- HIV-related diseases or living conditions)
* To evaluate theproportion of subjects with a pejorative event at 60 months of follow-up (recurrent or serious falls, emergency department visit, unscheduled hospitalization, institutionalization, loss of one point on the IADL scale or death)
* To evaluate the association between baseline frailty status and early / long-term pejorative events incidence
* Association between baseline evaluation of frailty and pejorative events incidence during the 60 months of follow-up.
* Transition between frail or non frail status during the 60 months of follow-up
* To assess the prevalence of sarcopenia and osteoporosis
* To describe study population including :

  * Demographic characteristics
  * HIV medical history and antiretroviral therapy
  * Comorbidities, polymedication and evaluation of drug-drug interactions
  * Mental Health, quality of life, socioeconomic status
  * Healthcare use and additional care implementation (nursing, physical therapy, home care services, …)
* Assessment of Inflammatory and Immunosenescence biomarkers at Baseline
* Anthropologic substudy about HIV and polypathologies management
* Focus on COVID-19 with clinical questionnaire, self-administrated questionnaire, SARS CoV2 serology and biobank (serum library)

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 70 years and older
* HIV-1 infection
* Antiretroviral therapy for at least 12 months
* Free and signed informed consent (article L1122-1-1-1 of the French Public Health Code)
* Person affiliated or benefiting from a social security scheme -

Exclusion Criteria:

* Participation in another research study excluding participation in other studies
* Person under legal protection or deprived of liberty by a judicial or administrative decision
* Isolated HIV-2 infection
* Life expectancy of less than 6 months

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 512 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2021-06-22 (Actual); Study Completion 2024-06-22 (Estimated)

PRIMARY OUTCOMES:
Proportion of frail patients at baseline | 12 months
  Proportion of patients classified as frail according to Fried at Baseline

SECONDARY OUTCOMES:
Proportion of frail subjects at M12, M24, M36, M48 and M60 | 60 months
  Proportion of frail subjects at M12, M24, M36, M48 and M60 according to Fried
Correlation between Baseline frailty status and early pejorative events incidence | 12 months
  Measure of association between frailty status and the existence of adverse health events (composite criterion defined by the existence of severe or repeated falls, use of emergency services, unscheduled hospitalization, institutionalization, loss of 1 point on the ADL scale, or death in the last 12 months)
Correlation between Baseline frailty status and long terme pejorative events incidence | 60 months
  Measure of association between frailty status and the existence of adverse health events (composite criterion defined by the existence of severe or repeated falls, use of emergency services, unscheduled hospitalization, institutionalization, loss of an ADL score, or death over the entire follow-up period to 60 months)
Transition between frail and non-frail status during 5 years of follow up | 60 months
  Evolution of the Fragility phenotype with estimation of the number of transitions from fragile to pre-fragile or robust status and the number of transitions from robust and pre-fragile status to fragile status.
Proportion of frail subjects accoding different frailty scores | 60 months
  Proportion of frail subjects according to different frailty indexes or scores : Fried, Cumulative Health deficits Index, French HAS score, VACS Index

CONTACTS AND LOCATIONS:
Overall Officials: Clotilde ALLAVENA, Principal Investigator — Infectious Diseases - CHU Nantes- France; Laurence MEYER, Principal Investigator — INSERM CESP - France; Hubert BLAIN, Principal Investigator — Geriatric Department - CHU Montpellier - France; Alain MAKINSON, Principal Investigator — Infectious Diseases - CHU Montpellier- France; Laurence SLAMA, Principal Investigator — Infectious Diseases - Hôtel Dieu Hospital Paris- France
Locations (1):
- Service de Maladies Infectieuses, CHU Hôtel-Dieu, Nantes, France

REFERENCES:
- [Derived] Sambou C, Pourette D, Debeaudrap P, Slama L, Katlama C, Cazanave C, Bonnet F, Meyer L, Allavena C. The burden of secrecy in the management of multimorbidity in older people living with HIV aged 70 and over. AIDS Care. 2024 Aug;36(8):1094-1101. doi: 10.1080/09540121.2024.2372723. Epub 2024 Jul 8. PMID 38976641